CLINICAL TRIAL: NCT02657226
Title: Association Between Intensive Monitoring of Renal Function and Outcomes in Critically Ill Patients
Brief Title: Intensive Monitoring of Renal Function
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: C. R. Bard (Industry)
Responsible Party: Principal Investigator, John Kellum, Director, Center for Critical Care Nephrology; Professor, Critical Care Medicine, University of Pittsburgh
Other Study IDs: PRO14120283
Record Dates: First submitted 2015-09-29; First posted 2016-01-15 (Estimated); Results first posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Intensive Monitoring of Renal Function; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intensive Monitoring of Renal Function: Urine output measurements recorded at least every 2 hours within the first 48 hours of ICU admission and serum creatinine measurements recorded daily for 3 days following ICU admission.
- Less-Intensive Monitoring of Renal Function: Urine output measurements with gaps of more than 3 hours recorded during the first 48 hours of ICU admission and fewer than 3 days of serum creatinine measurements after ICU admission.

SUMMARY:
This study aims to examine the association between monitoring (Intensive and non-intensive) of renal function (urine output, serum creatinine) and outcomes among critically ill patients such as Acute Kidney Injury (AKI) and mortality.

DETAILED DESCRIPTION:
Intensive monitoring of renal function provides an early opportunity to modify or attenuate certain risk factors (e.g., nephrotoxin exposure) for AKI. Intensive monitoring of urine output (UO) provides a real-time continuous assessment of renal function in the ICU. However, the association between intensive monitoring and less-intensive monitoring of urine output, with or without close monitoring of serum creatinine (sCr), on susceptibility to AKI and outcomes from AKI are unknown. Our preliminary data indicates that intensive monitoring of UO is associated with lower hospital mortality as compared to less-intensive monitoring for patients that develop AKI. If intensive monitoring of renal function is associated with lower risk of AKI and improved outcomes from AKI, then such monitoring techniques could be widely used in hospitalized patients including non-intensive care settings to either prevent AKI or progression of AKI.

Therefore, this observational retrospective cohort study aims to compare the outcomes of patients undergoing intensive monitoring of renal function (UO and/or sCr) with those of patients undergoing less intensive monitoring. Outcomes will include mortality within 30 days of ICU admission among critically ill patients with and without AKI. Development of severe AKI within 7 days of ICU admission and fluid overload on any ICU day in patients who develop severe AKI (KDIGO stage 3) will also be assessed.

This study will utilize a large, heterogeneous cohort (n=~54,800) of critically ill patients admitted to the ICU over 8 year period at the University of Pittsburgh Medical Center. The study population will consist of patients who receive intensive monitoring of UO (defined as measured at least every 2 hours within the first 48 hours of ICU admission) and strict creatinine measurement (defined as at least daily). Patients who fail to meet criteria for intensive monitoring will be controls (less-intensive monitoring group). AKI will be diagnosed according to the KDIGO stage 1-3 criteria over a 7-day period. Mortality at 30-days from ICU admission will be ascertained using the social security death master file. In order to account for indication bias, a propensity score for intensive monitoring will be built using various risk factors. Risk and severity of illness-adjusted estimates will be generated for susceptibility to AKI and mortality from AKI between intensive and less-intensive monitoring groups.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patient admitted to ICU
* Required vasopressor support or mechanical ventilation in the 24 hours from ICU admission

Exclusion Criteria:

* History of chronic dialysis and/or renal transplant
* Baseline serum creatinine >= 4 mg/dl
* Insufficient data to determine AKI stage in the 7 days from ICU admission
* Died within 48 hours from ICU admission
* ICU duration <2880 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted at the University of Pittsburgh Medical Center ICU or hospital.
Sampling Method: Non-Probability Sample
Enrollment: 15724 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2017-05 (Actual)

REFERENCES:
- [Result] Jin K, Murugan R, Sileanu FE, Foldes E, Priyanka P, Clermont G, Kellum JA. Intensive Monitoring of Urine Output Is Associated With Increased Detection of Acute Kidney Injury and Improved Outcomes. Chest. 2017 Nov;152(5):972-979. doi: 10.1016/j.chest.2017.05.011. Epub 2017 May 17. PMID 28527880
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/28527880

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an observational study. Hence, no prospective enrollment was performed. Collected data was analysed on patients meeting inclusion criteria for the study periof from year 2000 to 2008.
Groups:
- Study Population Undergoing Urine Output and Serum Creatinine: We stratified patients into two overlapping cohorts: those who received UO monitoring and those who received SC monitoring. We further subdivided each cohort into an intensive monitoring group and a less intensive monitoring group. UO intensive monitoring was defined as hourly recordings and no gaps of > 3 hours for the initial 48 hours after ICU admission, whereas less intensive UO monitoring was defined as patients not meeting intensive monitoring criteria regardless of UO information in the 7 days following ICU admission. SC intensive monitoring was defined as having 3 calendar days of SC data (at least one measure per day) after ICU admission, whereas less intensive SC monitoring was defined as patients not meeting intensive monitoring criteria regardless of SC monitoring availability in the 7 days following ICU admission.
Period: Overall Study
Arm/Group | Study Population Undergoing Urine Output and Serum Creatinine
Started | 15724
Completed (Total study population 15724.Patients were observed using different criteria of monitoring.) | 15724
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Population Undergoing Urine Output and Serum Creatinine
Number analyzed (Participants) | 15724
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [48 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6796
  Male | 8928
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American | 1164
  Race: White | 12276
  Race: Other | 2284
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15724

OUTCOME MEASURES:

1. Primary Outcome: Detection of Acute Kidney Injury (AKI)
Description: We classified AKI according to the maximum Kidney Disease Improving Global Outcomes criteria met during the 7 days after ICU admission using both SC and UO criteria. Admission creatinine levels were the first creatinine value recorded for the index hospital admission. Reference creatinine level was taken as the baseline creatinine level when available; otherwise, it was the lowest between admission creatinine level or creatinine level recorded in the 24 hours following ICU admission estimated using MDRD equation. For all analyses, we used moderate to severe AKI defined as stage 2-3. For UO criteria, at least every 6 hours data was required to stage AKI regardless of whether the patient had intensive or nonintensive UO monitoring overall.Odds ratio were measured between two groups.Odds ratios were determined using multivariable models for intensive vs non-intensive UO and between intensive vs non-intensive creatinine monitoring groups.
Time Frame: 7 days from ICU admission
Population: All patients receiving UO or SC monitoring
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Groups:
- Intensive vs Non-Intensive UO Monitoring; Intensive vs Non-Intensive SC Monitoring: We stratified patients into two overlapping cohorts: those who received UO monitoring and those who received SC monitoring. We further subdivided each cohort into an intensive monitoring group and a less intensive monitoring group. UO intensive monitoring was defined as hourly recordings and no gaps of > 3 hours for the initial 48 hours after ICU admission, whereas less intensive UO monitoring was defined as patients not meeting intensive monitoring criteria regardless of UO information in the 7 days following ICU admission. SC intensive monitoring was defined as having 3 calendar days of SC data (at least one measure per day) after ICU admission, whereas less intensive SC monitoring was defined as patients not meeting intensive monitoring criteria regardless of SC monitoring availability in the 7 days following ICU admission.
Arm/Group | Intensive vs Non-Intensive UO Monitoring | Intensive vs Non-Intensive SC Monitoring
Number analyzed (Participants) | 15724 | 15724
Odds Ratio
  Intensive monitoring urine output | 1.22 [1.11 to 1.35] | 1.22 [1.11 to 1.35]
  Intensive monitoring serum creatinine | 1.11 [1.00 to 1.24] | 1.11 [1.00 to 1.24]

2. Secondary Outcome: Mortality
Description: Hazard Ratios were measured to detect the risk of mortality at 30 days from ICU admission.
Time Frame: 30 days
Population: Intensive monitoring by urine output and serum creatinine among AKI population is reported.
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Study Population Undergoing Urine Output and Serum Creatinine
Number analyzed (Participants) | 15724
Hazard Ratio
  Intensive monitoring Urine Output | 0.90 [0.81 to 0.99]
  Intensive monitoring Serum Creatinine | 1.10 [0.98 to 1.24]

3. Secondary Outcome: Length of Stay in ICU
Description: Patients with and without AKI were compared among urine output group for duration of stay in ICU and hospital.
Time Frame: 30 days
Population: Median (Inter-Quartile Range) were reported.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Study Population Undergoing Urine Output and Serum Creatinine
Number analyzed (Participants) | 15724
days
  Uo Monitoring AKI | 8 [5 to 15]
  UO Monitoring No AKI | 5 [4 to 10]

4. Secondary Outcome: Hospital Length of Stay
Description: Hospital length of Stay was measured among urine output group and reported as median (Inter-Quartile Range).
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Study Population Undergoing Urine Output and Serum Creatinine
Number analyzed (Participants) | 15724
days
  UO Monitoring AKI | 17 [11 to 29]
  UO Monitoring no AKI | 14 [9 to 24]

ADVERSE EVENTS:
Description: This is a retrospective study. Adverse event reporting is not applicable.
Arm/Group | Study Population Undergoing Urine Output and Serum Creatinine
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This is a retrospective observational study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No